CLINICAL TRIAL: NCT06332261
Title: Standardized Assessment in Depression Treatment in Routine Psychiatric Services: a Retrospective Medical Record Review
Brief Title: Standardized Assessment in Depression Treatment in Routine Psychiatric Services
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Benjamin Bohman, Associate professor, Karolinska Institutet
Other Study IDs: 2024-BB-01
Record Dates: First submitted 2024-03-12; First posted 2024-03-27 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate current practices in depression treatment in psychiatric services in Stockholm, Sweden.

The main questions it aims to answer are:

* Are current practices consistent with local clinical guidelines in terms of standardized assessment and the treatments provided?
* What are the present conditions for implementing measurement-based care in depression treatment in this setting?

Data will be collected retrospectively from medical records of patients having received psychological or pharmacological treatment for depression from 2020 to 2023. Frequency of standardized assessments (not scores) using the Montgomery-Åsberg Depression Rating Scale, the Montgomery-Åsberg Depression Rating Scale-Self Assessment, and the Patient Health Questionnaire-9 is collected, together with information on patient, clinician, and treatment characteristics.

DETAILED DESCRIPTION:
Measurement-based care (MBC) refers to assessing outcomes prior to and during treatment with the purpose of providing a basis for treatment decisions and planning as treatment progresses (Lewis et al., 2019). MBC typically involves routine outcome monitoring on a session-to-session basis and clinical support tools to aid in the treatment process (Scott & Lewis, 2015; Trivedi, 2020). Research shows that MBC improves outcomes om symptom measures and reduces dropout as compared to treatment as usual without MBC (de Jong et al., 2021; Rognstad et al., 2023). Central to MBC is the frequent and systematic administration of outcome measures.

In public psychiatric services in Stockholm, Sweden, local clinical guidelines of the assessment and treatment of depression have been developed (Region Stockholm, 2021). These guidelines specify what psychological and pharmacological treatments to use, and at what time intervals assessment of outcomes should be conducted, and what measures to use. However, adherence to these guidelines in clinicians have not been evaluated; thus, it is not known to what extent the guidelines are properly implemented and what the present conditions are for introducing MBC in depression treatment in this setting.

Aims and research questions

A first aim of this study is to evaluate current practices in depression treatment in public psychiatric services in Stockholm. A second aim is to assess to what extent these practices adhere to local clinical guidelines, and if practices vary according to patient, clinician, and treatment characteristics. A third aim is to assess the present conditions for implementing MBC in depression treatment in this setting. The second aim provides valuable information for future initiatives of improving the conditions for implementing MBC in routine clinical practice settings. Research questions include:

1. Are current practices consistent with local clinical guidelines in terms of standardized assessment and the treatments provided?
2. Do current practices vary with patient, clinician, and treatment characteristics?
3. What are the present conditions for implementing MBC in depression treatment in this setting?

Design and procedure

This observational study employs a retrospective medical record review design. Medical records of patients initiating and completing treatment for major depression disorder between 1 January 2020 and 30 September 2023 at five general psychiatric clinics within public psychiatric outpatient services in Stockholm, Sweden are included. Specialized staff in this setting extract data on the frequency of standardized assessment, and patient, therapist, and treatment characteristics. Assessment points include at pre and post treatment as well as at specific points during treatment as specified in the local clinical guidelines.

Participants

Patients aged 18 years or older with major depressive disorder who have received psychological or pharmacological treatment.

Assessment

Frequency of standardized assessments (not scores) using the clinician-administered Montgomery-Åsberg Depression Rating Scale (MADRS; Montgomery & Åsberg, 1979), the self-reported Montgomery-Åsberg Depression Rating Scale-Self Assessment (MADRS-S; Svanborg & Åsberg, 2001), and the self-reported Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001) are collected. In addition, data are collected on patient characteristics (age, gender), clinician characteristics (age, gender, profession), and treatment characteristics, including clinic, type of treatment (psychological, pharmacological), type of psychological treatment (e.g., cognitive-behavioral, psychodynamic), type of pharmacological treatment (e.g., selective serotonin reuptake inhibitors), and treatment duration. The primary outcome measure is adherence to local clinical guidelines considering frequency of standardized assessments using the MADRS. Information identifying patients or clinicians is not collected.

Data analysis

Data on adherence of frequency of standardized assessments are examined using descriptive statistics. Group differences on categorical variables are investigated using chi-square tests or Kruskal-Wallis tests, and group differences on continuous variables are analyzed using multilevel modeling, taking account the nested data structure of patients and clinicians within clinics.

References

de Jong, K., Conijn, J. M., Gallagher, R. A. V., Reshetnikova, A. S., Heij, M., & Lutz, M. C. (2021). Using progress feedback to improve outcomes and reduce drop-out, treatment duration, and deterioration: a multilevel meta-analysis. Clinical Psychology Review, 85.

Kroenke, K., Spitzer, R. L., & Williams, J. B. (2001). The PHQ-9: validity of a brief depression severity measure. Journal of General Internal Medicine, 16(9), 606-13.

Lewis, C. C., Boyd, M., Puspitasari, A., Navarro, E., Howard, J., Kassab, H., Hoffman, M., Scott, K., Lyon, A., Douglas, S., Simon, G., & Kroenke, K. (2019). Implementing measurement-based care in behavioral health: a review. JAMA Psychiatry, 76(3), 324-35.

Montgomery, SA, & Åsberg, M. (1979). A new depression scale designed to be sensitive to change. British Journal of Psychiatry, 134, 382-9.

Region Stockholm (2021). Assessment and treatment of major depressive disorder. [Vårdprocesskarta för depression]. Region Stockholm, Stockholm, Sweden. Unpublished document.

Rognstad, K., Wentzel-Larsen, T., Neumer, S. P., & Kjøbli, J. (2023). A systematic review and meta-analysis of measurement feedback systems in treatment for common mental health disorders. Administration and Policy in Mental Health, 50(2), 269-82.

Scott, K., & Lewis, C. C. (2015). Using measurement-based care to enhance any treatment. Cognitive and Behavioral Practice, 22(1).

Svanborg, P., & Åsberg, M. (2001). A comparison between the Beck Depression Inventory (BDI) and the self-rating version of the Montgomery Asberg Depression Rating Scale (MADRS). Journal of Affective Disorders, 64, 203-16.

Trivedi, M. H. (2020). How can measurement-based care help improve treatment outcomes for major depressive disorder in primary care? Journal of Clinical Psychiatry, 81(2).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Principal diagnosis of major depressive disorder
* Psychological or pharmacological treatment initiated and completed between 1 January 2020 and 30 September 2023 at one of five general psychiatric clinics within public psychiatric outpatient services in Stockholm, Sweden

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of 18 years of age or older with a principal diagnosis of major depressive disorder who have initiated and completed psychological or pharmacological treatment between 1 January 2020 and 30 September 2023 at one of five general psychiatric clinics within public psychiatric outpatient services in Stockholm, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 2173 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale | Through study completion, an average of 1 year
  Ten-item clinician-administered measure of depressive symptoms

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale-Self Assessment | Through study completion, an average of 1 year
  Nine-item self-report version of the Montgomery-Åsberg Depression Rating Scale
The Patient Health Questionnaire-9 | Through study completion, an average of 1 year
  Nine-item self-report measure of depressive symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm Health Care Services, Region Stockholm, Stockholm, Sweden